CLINICAL TRIAL: NCT04619368
Title: Post-intensive Care Follow-up of Patients Hospitalized for an Acute Respiratory Distress Syndrome (ARDS) Caused by SARS-CoV-2 (COVID-19)
Brief Title: Post-intensive Care Follow-up of Patients Hospitalized for an Acute Respiratory Distress Syndrome Caused by COVID-19
Acronym: RE-CoV-ERY
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0219
Record Dates: First submitted 2020-11-03; First posted 2020-11-06 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Human ARDS; Coronavirus Infection
Keywords: Post-intensive care Syndrome; Acute Respiratory Distress Syndrome; quality of life; intensive care unit; PTSD; follow-up after ICU; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections; postintensive care syndrome; Stress Disorders, Post-Traumatic; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Follow up calls — The follow-up will consist in phone call with an intensive care doctor. These visits would be the opportunity to screen the complications after intensive-care with, find solutions to cure them or decrease their impact on patient's life to improve quality of life and prevent the post-traumatic syndrome disorder PTSD. A review would be sent to the patients' General Practitioners at the end of each visit.

SUMMARY:
For the last years, studies have described the " Post-intensive care Syndrome " (PICS), which consists in alteration of quality of life, cognition, autonomy and psychological disorders within the months after intensive-care. Patients with COVID-19 in intensive care units are at high risks to develop PICS.

The primary objective is to analyse the incidence of the post-traumatic stress disorder at 12 months after intensive-care for a COVID-19 Acute Respiratory Distress Syndrome (ARDS).

DETAILED DESCRIPTION:
Many studies have showed that ARDS survivors keep, even a long time after hospitalization, a functional respiratory disability, resulting on one hand from impaired diffusion of carbon monoxide, and on the other hand from a muscular weakness. Indeed, 67% of patients ventilated more than 10 days have a neuromyopathy whose recovery is uncertain.

Beside this, Long-term quality of life is worse than in general population, due in particular to depressive and anxiety disorders such as post-traumatic syndrome disorder with a prevalence around 22% after one year.

The follow-up will consist in phone call with an intensive care doctor. These visits would be the opportunity to screen the complications after intensive-care with, find solutions to cure them or decrease their impact on patient's life to improve quality of life and prevent the post-traumatic syndrome disorder PTSD. A review would be sent to the patients' General Practitioners at the end of each visit.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* hospitalized in intensive care of the CHU anesthesia-intensive care unit (Rangueil, URM, Neurosurgery)
* intubated and ventilated
* supported for an ARDS according to the Berlin criteria (PaO2 / FiO2 ratio <300 mmHg)
* with an rt-PCR positive to SARS-CoV-2
* affiliated to the french social security

Exclusion Criteria:

* minor patient
* patient under protective measure
* ARDS in the pandemic context but rt-PCR negative to SARS-CoV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cohort of all COVID patients who went out alive from intensive care
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Post-traumatic Stress Disorder (PTSD) with the Post-traumatic Checklist-5 (PCL-5) 12 months after intensive-care | month 12
  Incidence of Post-traumatic Stress Disorder (PTSD) with the Post-traumatic Checklist-5 (PCL-5) 12 months after intensive-care

SECONDARY OUTCOMES:
psychological disorders measured by QIDS | Month 3
  psychological disorders measured by QIDS, Quick Inventory of Depressive Symptomatology. results from 0 to 27; 27 is the higher score of depressive symptoms
psychological disorders measured by STAI-YA | Month 3
  psychological disorders measured by STAI-YA, State Trait Inventory Anxiety. Results from 20 to 80. 80 is the higher score of anxiety
psychological disorders measured by QIDS | Month 6
  psychological disorders measured by QIDS : Quick Inventory of Depressive Symptomatology. results from 0 to 27; 27 is the higher score of depressive symptoms
psychological disorders measured by STAI-YA | Month 6
  psychological disorders measured by STAI-YA, State Trait Inventory Anxiety. Results from 20 to 80. 80 is the higher score of anxiety
psychological disorders measured by QIDS | Month 12
  psychological disorders measured by QIDS, Quick Inventory of Depressive Symptomatology. results from 0 to 27; 27 is the higher score of depressive symptoms
psychological disorders measured by STAI-YA | Month 12
  psychological disorders measured by STAI-YA, State Trait Inventory Anxiety. Results from 20 to 80. 80 is the higher score of anxiety
quality of life by EQL-5 | Month 3
  Quality of life measured by European Quality of Life -5 scale (overall satisfaction of Europeans concerning different aspects of life) higher score is higher quality of life
quality of life by EQL-5 | Month 6
  Quality of life measured by European Quality of Life -5 scale (overall satisfaction of Europeans concerning different aspects of life), higher score is higher quality of life
quality of life by EQL-5 | Month 12
  Quality of life measured by European Quality of Life -5 scale (overall satisfaction of Europeans concerning different aspects of life), higher score is higher quality of life
nutritional status | Month 3
  nutritional status measured by Nutritional Risk Screening 2002
nutritional status | Month 6
  nutritional status measured by Nutritional Risk Screening 2002
nutritional status | Month 12
  nutritional status measured by Nutritional Risk Screening 2002

CONTACTS AND LOCATIONS:
Overall Officials: Fanny BOUNES, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided